CLINICAL TRIAL: NCT07087600
Title: Immediate Effects on Ventilatory Morphofunctional Pattern and Cardiorespiratory Safety During Automatic Body Lateralization Therapy in Critically Ill Patients: A Quasi-Experimental Study
Brief Title: Immediate Effects of Automatic Lateralization in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other); Coordination for the Improvement of Higher Education Personnel (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Shirley Lima Campos, Principal Researcher, University of Pernambuco
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70188523.0.0000.5200
Record Dates: First submitted 2024-08-16; First posted 2025-07-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Intensive Care Units
Keywords: Automatic lateralization therapy; Critical illness; Continuous lateral rotation; Electrical impedance tomography
MeSH Terms: conditions — Critical Illness | interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental, before-and-after study, and contains a single group, in which the group itself is the control. There will be a comparison before, during and after the intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic lateralization therapy (Active Comparator): Participants will undergo automatic lateral positioning using a motorized bed programmed to alternate angles of 0°, 15°, and 30°, switching sides continuously.
  Interventions: Other: Automatic lateralization therapy
- Supine position (Active Comparator): Participants will remain in supine position with 30° head elevation. No lateralization therapy is applied.
  Interventions: Other: Supine Positioning

INTERVENTIONS:
Other: Automatic lateralization therapy — Program the bed to vary angle and time continuously during the intervention
  Other Names: Continuous lateral positioning; kinetic therapy; automated lateral rotation therapy
  Arms: Automatic lateralization therapy
Other: Supine Positioning — In this intervention, participants will be positioned in the supine position with the head of the bed elevated at 30°
  Other Names: Supine; Semi-recumbent position; Recumbent position; Dorsal decubitus; Conventional supine care
  Arms: Supine position

SUMMARY:
New devices have been used in intensive care to optimize respiratory function in critically ill patients, such as automatic lateralization therapy. However, the times and angles used vary widely, and there is no clear evidence of cardiovascular safety and immediate effects, which represents a gap in the literature. This quasi-experimental study aims to evaluate the imediact efficacy and cardiorespiratory safety of automatic lateralization therapy in critically ill patients under invasive mechanical ventilation. The primary outcomes include changes in ventilation distribution and end-expiratory impedance variation. Secondary outcomes include respiratory mechanics, vital signs, and adverse events.

DETAILED DESCRIPTION:
Introduction: Electrical impedance tomography (EIT) enables real-time imaging of lung ventilation, guiding interventions such as automatic lateralization therapy. Despite its potential, evidence about immediate effects and safety is limited.

Objective: To evaluate the imediact cardiorespiratory efficacy and safety of automatic lateralization therapy in critically ill patients.

Method: Quasi-experimental, non-randomized, two-arm study. Participants aged ≥18 years, intubated and clinically stable, will undergo both interventions.

Interventions:

* Arm 1: Supine position with head elevated at 30°.
* Arm 2: Automatic lateralization therapy using programmable bed angles (0°, 15°, and 30°), alternating sides.

Outcomes: Ventilation distribution, impedance variation (ΔZ, ΔEELZ), respiratory mechanics, adverse events, and vital signs will be measured.

Ethical approval has been granted (CAAE 70188523.0.0000.5200). Informed consent will be obtained from legal guardians.

ELIGIBILITY:
Inclusion criteria:

* Volunteers aged 18 or over;
* Of both sexes;
* Breathing through an orotracheal tube;
* With respiratory and hemodynamic stability.

Exclusion criteria:

* Patients with contraindications to change of position;
* Acute spinal cord injury;
* Unstable fractures and signs of intracranial hypertension;
* Pregnant women;
* Immediate postoperative period of thoracic, orthopedic and abdominal surgeries;
* Use of drains;
* Grade III obesity (BMI > 40 kg/m2);
* Suspected pulmonary thromboembolism;
* Agitation and active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Electrical impedance tomography (EIT): End-Expiratory Electrical Impedance Variation (ΔEELZ) | In the 5 minutes of each angulation, totaling 15 minutes in the unilateral morphofunctional pattern or 20 minutes in the bilateral morphofunctional pattern.
  Represents the change in regional pulmonary aeration between the pre- and post-intervention moments.
Electrical impedance tomography (EIT): Ventilation Distribution Variation (ΔZ) | In the 5 minutes of each angulation, totaling 15 minutes in the unilateral morphofunctional pattern or 20 minutes in the bilateral morphofunctional pattern.
  Represents the change in ventilation distribution before and after the intervention.

SECONDARY OUTCOMES:
Adverse events | In the 5 minutes of each angulation, totaling 15 minutes in the unilateral morphofunctional pattern or 20 minutes in the bilateral morphofunctional pattern.
  Monitoring of serious and non-serious adverse events associated with the intervention through an adapted adverse event form
Respiratory Mechanics | In the 5 minutes of each angulation, totaling 15 minutes in the unilateral morphofunctional pattern or 20 minutes in the bilateral morphofunctional pattern.
  Data provided through the mechanical ventilator and from inspiratory and expiratory pause maneuvers
Vital signs | In the 5 minutes of each angulation, totaling 15 minutes in the unilateral morphofunctional pattern or 20 minutes in the bilateral morphofunctional pattern.
  Viewed on the multiparameter monitor

OTHER OUTCOMES:
Lung morphofunctional pattern | In the 5 minutes of each angulation, totaling 15 minutes in the unilateral morphofunctional pattern or 20 minutes in the bilateral morphofunctional pattern.
  Type of pattern of lung alteration observed by functional electrical impedance tomography image (preserved, unilateral involvement, unilateral dorsal, bilateral, bilateral dorsal).

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Lima Campos, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Hospital Geral Otávio de Freitas, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, anonymized data will be made available for scientific use, as:
  * Participant characteristics (age, gender)
  * Clinical measurements (blood pressure, heart rate)
  * Medical history
  * Clinical laboratory results
  * Adverse events (hemodynamic and respiratory instability, interruptions)
  * Details of treatment received
Supporting Information: Study Protocol, SAP, ICF
Time Frame: End of trial
Access Criteria: Individual participant data (IPD) access will be granted by the PI after request review for approval via email. It will be shared with researchers and general public of interest on the subject for descriptive analyses related to our sample medical and clinical characteristics. A committee of researchers will be in charge of discussing the request before approving the access.

REFERENCES:
- [Background] American Association for Respiratory Care. AARC Clinical Practice Guidelines. Endotracheal suctioning of mechanically ventilated patients with artificial airways 2010. Respir Care. 2010 Jun;55(6):758-64. PMID 20507660
- [Background] Maclin VM, Radwanska E, Binor Z, Dmowski WP. Progesterone:estradiol ratios at implantation in ongoing pregnancies, abortions, and nonconception cycles resulting from ovulation induction. Fertil Steril. 1990 Aug;54(2):238-44. doi: 10.1016/s0015-0282(16)53696-6. PMID 2379624
- [Background] Doering LV. The effect of positioning on hemodynamics and gas exchange in the critically ill: a review. Am J Crit Care. 1993 May;2(3):208-16. PMID 8364672
- [Background] Doerschug KC, Schmidt GA. Intensive care ultrasound: III. Lung and pleural ultrasound for the intensivist. Ann Am Thorac Soc. 2013 Dec;10(6):708-12. doi: 10.1513/AnnalsATS.201308-288OT. No abstract available. PMID 24364779
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Hassan AA, Evrensel CA, Krumpe PE. Clearance of viscoelastic mucus simulant with airflow in a rectangular channel, an experimental study. Technol Health Care. 2006;14(1):1-11. PMID 16556959
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Kang SY, DiStefano MJ, Yehia F, Koszalka MV, Padula WV. Critical Care Beds With Continuous Lateral Rotation Therapy to Prevent Ventilator-Associated Pneumonia and Hospital-Acquired Pressure Injury: A Cost-effectiveness Analysis. J Patient Saf. 2021 Mar 1;17(2):149-155. doi: 10.1097/PTS.0000000000000582. PMID 30896557
- [Background] Molina FJ, Rivera PT, Cardona A, Restrepo DC, Monroy O, Rodas D, Barrientos JG. Adverse events in critical care: Search and active detection through the Trigger Tool. World J Crit Care Med. 2018 Feb 4;7(1):9-15. doi: 10.5492/wjccm.v7.i1.9. eCollection 2018 Feb 4. PMID 29430403
- [Background] Politi S, Aloisi A Jr, Bartoli V, Guglietta A, Magnifica F. Infrared Thermography Images Acquisition for a Technical Perspective in Screening and Diagnostic Processes: Protocol Standardized Acquisition. Cureus. 2021 Nov 27;13(11):e19931. doi: 10.7759/cureus.19931. eCollection 2021 Nov. PMID 34976527
- [Background] Roldan R, Rodriguez S, Barriga F, Tucci M, Victor M, Alcala G, Villamonte R, Suarez-Sipmann F, Amato M, Brochard L, Tusman G. Sequential lateral positioning as a new lung recruitment maneuver: an exploratory study in early mechanically ventilated Covid-19 ARDS patients. Ann Intensive Care. 2022 Feb 12;12(1):13. doi: 10.1186/s13613-022-00988-9. PMID 35150355
- [Background] Staudinger T, Bojic A, Holzinger U, Meyer B, Rohwer M, Mallner F, Schellongowski P, Robak O, Laczika K, Frass M, Locker GJ. Continuous lateral rotation therapy to prevent ventilator-associated pneumonia. Crit Care Med. 2010 Feb;38(2):486-90. doi: 10.1097/CCM.0b013e3181bc8218. PMID 19789440
- [Background] Teasell R, Dittmer DK. Complications of immobilization and bed rest. Part 2: Other complications. Can Fam Physician. 1993 Jun;39:1440-2, 1445-6. PMID 8324412
- [Background] Volpe MS, Guimaraes FS, Morais CC. Airway Clearance Techniques for Mechanically Ventilated Patients: Insights for Optimization. Respir Care. 2020 Aug;65(8):1174-1188. doi: 10.4187/respcare.07904. PMID 32712584
- [Background] Wanless S, Aldridge M. Continuous lateral rotation therapy - a review. Nurs Crit Care. 2012 Jan-Feb;17(1):28-35. doi: 10.1111/j.1478-5153.2011.00458.x. Epub 2011 Jul 20. PMID 22229679
- See also: Multicare: cama articulável para cuidado intensivo — https://drive.google.com/file/d/1d5w2gER61YmaYc7Wn0vKFwyVFD6lw5pD/view?usp=sharing